CLINICAL TRIAL: NCT03852095
Title: Single Time Management for Seven Common Disease in Pediatric Traumatology. A Monocentric Prospective Study
Brief Title: Single Time Management Diseases in Pediatric Traumatology
Status: Completed | Type: Observational
Sponsor: Fondation Lenval (Other)
Responsible Party: Sponsor
Other Study IDs: 18-HPNCL-06
Record Dates: First submitted 2019-02-21; First posted 2019-02-22 (Actual); Last update posted 2019-07-19 (Actual); Status verified 2019-02

CONDITIONS: Fractures, Bone
Keywords: Pediatric, traumatology, hemarthrosis, ankle, knee,; buckle fracture, clavicle, sprains
MeSH Terms: conditions — Fractures, Bone; Hemarthrosis; Sprains and Strains

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- minor trauma: Child from 1 to 18 years old suffering an isolated minor trauma presenting at the hospital emergency services.
  Interventions: Other: minor trauma

INTERVENTIONS:
Other: minor trauma — following the management of the patient's fracture in the emergency department, the patients / parents are recalled 2 months (J60) after the visit to the emergency room, and are interviewed by following the pre-established interrogation form, which checks the good agreement of the patient. treatment performed with the given sheet and recommendations, and assesses the satisfaction.
  Other Names: medical recommendation sheet

SUMMARY:
A recent internal study evaluating the relevance of the visit to traumatology consultation in our establishment highlight that 49.3% of consultations were not relevant passages. The project consists of individualizing 5 to 6 pathologies and to create care sheets and patient sheets to be given to the care teams and patients when the pathology lends itself to it. The aim is to reduce the irrelevant passage rate during these consultations, which is the source of absence from iterative work for parents, collateral expenses (toll, parking), absence from school for the children, unjustified expenses and X-ray examination unnecessary most often.

DETAILED DESCRIPTION:
The Pediatric Orthopedics and Traumatology department proposes a reform of the care in Traumatology of the children in order to improve and homogenize the care for a better relevance of these.

A recent internal study (June 2018) evaluating the relevance of the visit to traumatology consultation in our establishment to highlight that 49.3% of consultations were not relevant passages (Benign diseases of sprained ankle type, muscular contusion or simple bone removals). Indeed, these specialist consultations are currently filled by pathologies of simple treatment that do not require medical follow-up (neither clinical nor radiological follow-up).

The project consists of individualizing 5 to 6 pathologies found in consultation recurrently which the scientific literature has established that their follow-up is not justified, and to create care sheets and patient sheets to be given to the care teams and patients when the pathology lends itself to it. These cards will include all the management of the pathology of the definition itself, including the treatment and expected outcomes.

The aim is to reduce the irrelevant passage rate during these consultations, which is the source of absence from iterative work for parents, collateral expenses (toll, parking), absence from school for the children, unjustified expenses and X-ray examination unnecessary most often.

The expected benefit is parental and child satisfaction, a time saving for the practitioner that he can reinvest in consultations for patients who are in fact a specialist opinion and a relative budget saving for the establishment.

The method of study of the decline of irrelevant consultations will be made by a systematic review of each reason for consultation over a period of 3 months after implementation of the cards and study of the percentage of irrelevant consultation over the same period. The objective pursued is a drop in attendance of at least 25% of consultations deemed irrelevant in Traumatology, associated with a satisfaction rate of parents greater than 90%.

ELIGIBILITY:
Inclusion Criteria:

* 0-18 years
* Positive diagnosis of elbow haemarthrosis, radial salter 1 fracture, fibula fracture 1 fracture, radial butter ball fracture, simple ankle sprain, simple knee sprain, fracture of the middle third of the clavicle .........
* No other associated anomaly

Exclusion Criteria:

* Refusal of the family ..............................................
* No understanding of the instructions ...............................
* Unaffiliated patient social security ..................................
* No French speaking .............

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Child from 1 to 18 years old suffering an isolated minor trauma presenting at the Lenval Foundation emergency services.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2018-11-02 (Actual); Primary Completion 2019-06-14 (Actual); Study Completion 2019-06-28 (Actual)

PRIMARY OUTCOMES:
Change of the number of patients routinely summoned to post-emergency trauma consultation | at 6 months
  decrease in the number of patients coming back for an unjustified consultation for these 4 pathologies by comparing the period from 6 months preceding the start of the protocol to a period of 6 months after starting the protocol.

SECONDARY OUTCOMES:
measurement of patient satisfaction | at 60 days after inclusion
  Call by phone the patient to measure the satisfaction by a standard questionnaire. the scale is composed of 7 closed questions on the satisfaction of care in emergencies, the follow-up of the patient by a city doctor. the answers are yes or no.
compliance of care | at 60 days after inclusion
  call by phone the patient to verify the good compliance of the care. The improvement of the care will be evaluated according to the number of patient treated for one of these pathologies having felt the need to consult another doctor / orthopedic surgeon that is envisaged by the protocol (in the days following emergency room consultation).

CONTACTS AND LOCATIONS:
Overall Officials: RAMPAL VIRGINIE, MD, Principal Investigator — Fondation Lenval - Nice Children Hospital CHU-Lenval
Locations (1):
- Fondation Lenval Hopitaux Pediatriques de Nice Chu Lenval, Nice, France